CLINICAL TRIAL: NCT06411600
Title: Bevacizumab Plus encoRAfenib-cetuximab in BRAF-V600E Mutated Metastatic Colorectal Cancer, a Phase II Study With a Safety lead-in Cohort, the BRAVE Trial
Brief Title: Combination Therapy for BRAF-V600E Metastatic CRCm
Acronym: BRAVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VHIO23001
Record Dates: First submitted 2024-04-24; First posted 2024-05-13 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Encorafenib; Cetuximab; Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — encorafenib; Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): The experimental arm in the BRAVE protocol involves the administration of a combination therapy consisting of encorafenib, cetuximab, and bevacizumab. This arm is designed to evaluate the efficacy and safety of this combination in patients with metastatic colorectal cancer harboring the BRAF-V600E mutation who have experienced disease progression after one or two prior chemotherapy regimens. The primary objective is to assess the antitumor activity of the combination therapy, with secondary objectives including safety and tolerability assessments, as well as evaluations of progression-free survival, overall survival, and patient-reported outcomes.
  Interventions: Drug: Encorafenib; Drug: Cetuximab; Drug: Bevacizumab
- Control arm (Active Comparator): The control arm in the BRAVE protocol involves standard-of-care treatment, which may include various chemotherapy regimens or targeted therapies typically used for metastatic colorectal cancer. In this arm, patients receive the standard treatment without the addition of encorafenib, cetuximab, or bevacizumab. The purpose of the control arm is to provide a reference point for comparing the efficacy and safety of the experimental combination therapy. Patients in this arm may also undergo similar assessments for tumor response, survival outcomes, and adverse events to facilitate comparison with the experimental arm.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Encorafenib — Encorafenib is administered orally at a daily dose of 300 mg, typically in the form of four 75 mg capsules taken together.
  Arms: Experimental arm
Drug: Cetuximab — Cetuximab is administered intravenously every two weeks at a dose of 500 mg/m².
  Arms: Experimental arm
Drug: Bevacizumab — Bevacizumab is administered intravenously every two weeks at a dose of 5 mg/kg.

SUMMARY:
The BRAVE is a phase II clinical trial aimed at evaluating the efficacy of the combination therapy of encorafenib, cetuximab, and bevacizumab in patients with metastatic colorectal cancer (CRC) harboring the BRAF-V600E mutation. This mutation is present in about 8-10% of CRC cases and is associated with poor prognosis and limited treatment options. The rationale behind this trial stems from preclinical studies suggesting that the overexpression and activation of vascular endothelial growth factor A (VEGFA) may contribute to resistance to BRAF inhibitors (BRAFi) in CRC. Thus, the trial hypothesizes that adding bevacizumab, an anti-angiogenic agent targeting VEGFA, to the combination of encorafenib and cetuximab may delay acquired resistance, leading to improved progression-free survival.

The primary objective of the BRAVE is to evaluate the antitumor activity of the encorafenib-cetuximab-bevacizumab combination in patients who have experienced disease progression after one or two chemotherapy regimens for BRAF V600E-mutant metastatic CRC. This activity will be assessed based on the confirmed progression-free survival rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

DETAILED DESCRIPTION:
Study Design: The study adopts a multicenter, open-label, phase II design. Patients with metastatic CRC harboring the BRAF-V600E mutation, who have experienced disease progression after one or two prior chemotherapy regimens, are eligible for enrollment. The treatment regimen consists of daily oral encorafenib (300 mg), biweekly intravenous cetuximab (500 mg/m2), and biweekly intravenous bevacizumab (5 mg/kg). Treatment will be administered in 28-day cycles until disease progression, unacceptable toxicity, consent withdrawal, initiation of other anticancer therapy, or death.

Secondary Objectives: Secondary objectives include evaluating the safety and tolerability of the combination therapy, assessing objective response rate, time to response, duration of response, overall survival, and patient-reported outcomes. Exploratory objectives involve evaluating potential biomarkers predictive of treatment response and resistance, as well as generating functional models to assess novel drug combinations targeting resistance mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Age ≥18 years at time of informed consent.
* Histologically- or cytologically-confirmed mCRC that is metastatic.
* Presence of BRAF V600E mutation in tumor tissue previously determined according to the guidelines of each center, any time point before the enrollment in the study.
* Microsatellite stability must be confirmed according to the guidelines of each center, any time point before the enrollment in the study.
* Eligible to receive cetuximab per locally approved label with regard to tumor RAS status, any time point before the enrollment in the study.
* Progression of disease after 1 or 2 prior regimens in the metastatic setting.
* Evidence of measurable or evaluable non-measurable disease per RECIST, v1.1.
* ECOG PS of 0 or 1.
* Adequate bone marrow function characterized by the following at screening:

  1. Absolute neutrophil count (ANC) ≥1.5 x 109/L
  2. Platelets ≥100 x 109/L
  3. Hemoglobin ≥9.0 g/dL (with or without blood transfusions).
* Adequate hepatic and renal function characterized by the following at screening:

  1. Serum total bilirubin ≤1.5 x upper limit of normal (ULN) and <2 mg/dL. Note: Total bilirubin >1.5 x ULN is allowed if direct (conjugated) ≤1.5 x ULN and indirect (unconjugated) bilirubin is ≤4.25 x ULN. Note: Participants with hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the Sponsor medical monitor.
  2. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 x ULN, or ≤5 x ULN in the presence of liver metastases.
  3. Adequate renal function defined by an estimated creatinine clearance ≥50 mL/min according to the Cockcroft Gault formula or by 24-hour urine collection for creatinine clearance, or according to local institutional standard method.
  4. Protein < 2+ on dipstick urinalysis or ≤ 1.0 g in a 24-hour urine collection. All patients with ≥2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.
  5. Adequate electrolytes, defined as serum potassium and magnesium levels within institutional normal limits.

Note: Replacement treatment to achieve adequate electrolytes will be allowed.

* Adequate cardiac function characterized by the following at screening:

  a.Mean triplicate QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤480 msec.
* Able to take oral medications.
* Highly effective contraception for both male and female subjects if the risk of conceptions exists during and at least up to 6 months after the last medication. See 10.4. Appendix 4.

Exclusion Criteria:

* Treatment with another investigational drug or participation in another investigational study at enrolment or within 30 days prior to enrolment.
* Patient unable to comply with the study protocol owing to psychological, social (lack of social support or social exclusion) or geographical reasons.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Cycle 1, Day 1.
* Evidence of bleeding diathesis or clinically significant coagulopathy (in the absence of therapeutic anticoagulation).
* Patients with history of pulmonary hemorrhage/hemoptysis (>1/2 teaspoon red blood) within 6 months prior to Cycle 1, Day 1.
* Known history of acute or chronic pancreatitis.
* Tumors with microsatellite instability or mismatch repair deficiency.
* History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention. (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months before the enrollment in the study.
* Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

  1. History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft [CABG], coronary angioplasty or stenting) ≤ 6 months prior to start of study treatment.
  2. Symptomatic congestive heart failure (i.e., Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality ≤ 6 months prior to start of study treatment, except atrial fibrillation and paroxysmal supraventricular tachycardia.
* Uncontrolled hypertension defined as persistent systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg despite current therapy.
* Impaired hepatic function, defined as Child-Pugh class B or C.
* Known history of human immunodeficiency virus (HIV), active hepatitis B virus (HBV) infection or active hepatitis C virus (HCV) infection. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients with past exposure to HBV are also eligible for the study provided they are negative for HBV DNA.
* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and the enrollment in the study.
* Subjects with leptomeningeal carcinomatosis.
* Impaired gastrointestinal (GI) function or disease that may significantly alter the absorption of encorafenib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).
* Concurrent or previous other malignancy within 5 years of study entry without Sponsor approval, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, or other noninvasive or indolent malignancy.
* History of thromboembolic or cerebrovascular events ≤ 6 months prior to starting study treatment, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis or pulmonary embolism.
* Knowledge of any other disease or medication that may interfere with study treatment.
* Known severe hypersensitivity reactions to monoclonal anti-bodies or BRAF inhibitors.
* Known hypersensitivity to any of encorafenib, cetuximab or bevacizumab-bvzr active ingredients or their excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Until disease progression, typically within a follow-up period of approximately 5 years.
  PFS will be evaluated by local radiologist/investigator assessment per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1). It refers to the duration from the start of treatment until disease progression or death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Throughout the study duration, that it will take 5 years
  ORR will be determined as the proportion of patients achieving a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.
Duration of Response (DOR) | Until disease progression, typically within a follow-up period of approximately 5 years.
  DOR is defined as the duration from the first radiographic evidence of response to the earliest documented disease progression or death due to underlying disease.
Disease Control Rate (DCR) | Throughout the study duration, that it will take 5 years
  The proportion of patients who achieve a complete response, partial response, or stable disease as the best overall response to treatment.
Electrocardiogram (ECG) Changes | During treatment (until disease progression) and up to 30 ± 2 days after the last dose.
  This outcome measure assesses changes in electrocardiogram (ECG) parameters in participants receiving treatment with encorafenib in combination with cetuximab and bevacizumab, as well as up to 30 ± 2 days after the last dose. ECG recordings will be analyzed for parameters such as QT interval duration, presence of arrhythmias, and other relevant ECG changes.
Incidence and Severity of Adverse Events | Until disease progression, typically within a follow-up period of approximately 5 years.
  This outcome measure assesses the occurrence and severity of adverse events experienced by participants during treatment with encorafenib in combination with cetuximab and bevacizumab, as well as up to 30 ± 2 days after the last dose. Adverse events will be categorized and graded according to standardized criteria (e.g., CTCAE version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Elez, MD PhD, Principal Investigator — Vall d'Hebron Institute of Oncology
Locations (1):
- Vall d'Hebron Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No